CLINICAL TRIAL: NCT07091578
Title: Assessing the Feasibility of School-Based Oral Health Programmes in Primary Schools in Saudi Arabia: A Pilot Study
Brief Title: Supervised Toothbrushing and Oral Health Education in Primary Schools in Saudi Arabia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatimah Alshehri (Other)
Collaborators: King Saud University (Other)
Responsible Party: Sponsor-Investigator, Fatimah Alshehri, Principal Investigator, King's College London
Organization: King's College London (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: LRS/DP-23/24-40999; 24/1240/IRB (Other: King Saud University)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries
Keywords: Dental Caries; Children; Toothbrushing; Oral Health Education; Primary Schools
MeSH Terms: conditions — Dental Caries | interventions — Health Education, Dental

STUDY DESIGN:
Intervention Model Description: This study employed a pilot study with three parallel groups. The study was carried out in three public primary schools in Riyadh, Saudi Arabia, for one calendar year. Each school is assigned to either supervised toothbrushing or oral health education with a 1:1:1 allocation ratio. Students, school staff, and dental professionals were actively involved in this study. Students were engaged in oral health programmes throughout the academic year, enabling a thorough evaluation of the interventions' impact on their oral health. School staff and dental professionals conducted the interventions; their feedback will be valuable in identifying facilitators and barriers to the implementation. This design provides useful insights into the barriers and facilitators of delivering oral health programmes in primary schools, allowing for testing programme feasibility before conducting larger-scale implementation in the future (Eldridge and Kerry, 2012).
Who Masked: Outcomes Assessor
Masking Description: This study adopted a single-blinded approach, with an assessor blinded to the interventions. Blinding was implemented by maintaining a clear separation of roles. The dental professionals delivering interventions were not involved in outcome assessments, and outcome assessors did not have access to information about the specific interventions received by participants. Once schools had been assigned to intervention groups, students, school staff, and the dental professionals delivering interventions were blinded due to the nature of the intervention. However, outcome assessors responsible for conducting dental examinations were blinded to participants' assigned intervention groups to minimise potential bias. Dentists acted as outcome assessors and performed baseline and follow-up dental examinations, whereas dental hygienists oversaw the interventions, including supervised toothbrushing and oral health education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Toothbrushing (Experimental): Children participated in a daily supervised toothbrushing programme conducted in school and received monthly oral health educational sessions by trained teachers and the dental team.
  Interventions: Behavioral: Supervised toothbrushing
- Oral Health Education (Active Comparator): Children received oral health education sessions in the classrooms provided by trained teachers and the dental team.
  Interventions: Behavioral: Oral Health Education

INTERVENTIONS:
Behavioral: Supervised toothbrushing — In supervised toothbrushing intervention, dental hygienists trained school staff, obtained consent forms, distributed the oral hygiene kits, and provided support and advice if needed. Teachers' training included guidelines for infection prevention and control, and toothbrushing in dry areas adapted from the Public Health England (PHD) toothbrushing programme toolkit. A dry toothbrushing model was employed. Toothbrushing sessions took place daily during regular school hours for one academic year. Each session lasted for approximately 10 minutes and occured after break time at 9:20 am. Oral hygiene kits that include soft toothbrushes and 1450ppm fluoridated toothpaste were disseminated every three months. Teachers and dental hygienists provided monthly oral health educational sessions to students during regular school time.
  Arms: Supervised Toothbrushing
Behavioral: Oral Health Education — In oral health education intervention, dental hygienists and school staff collaborated to educate students about oral health. Dental hygienists trained school staff to deliver this programme effectively and offer continued support and guidance to school staff during the programme implementation. An oral health education toolkit partly adapted from the PHE toothbrushing programme toolkit was provided to the school before the start of the programme. Educational materials including lectures, leaflets, and activities were dispensed monthly. Oral health education was conducted once a month during regular school hours in the classroom, and each session lasted for one hour. Students were provided with comprehensive knowledge about oral health, such as proper toothbrushing techniques, the importance of routine dental check-ups, and healthy nutrition. Moreover, toothbrushing kits that include soft toothbrushes and 1450ppm fluoridated toothpaste were distributed every three months.
  Arms: Oral Health Education

SUMMARY:
The goal of this pilot study is to assess the feasibility of implementing school-based oral health programmes including supervised toothbrushing and oral health education. The main questions it aims to answer are:

* Is it feasible to implement supervised toothbrushing and oral health education programmes in primary schools in Riyadh, Saudi Arabia?
* What are the facilitators and barriers to implementation regarding programme acceptance, participation of school staff, and adherence to the supervision guidelines?
* How do these programmes influence children's self-reported oral health status, risk behaviours, and quality of life during the study period?
* What is the effect of these programmes on dental caries incidence, plaque and gingival bleeding scores over a one-year follow-up?

Participants will:

* Take part in either a supervised toothbrushing programme or an oral health education programme.
* Undergo dental examinations at baseline and after one year of follow-up to assess changes in dental caries, and plaque and gingival bleeding scores.

DETAILED DESCRIPTION:
Dental caries is one of the most widespread oral health diseases affecting populations worldwide, including Saudi Arabia. Several studies assessing dental caries prevalence in Saudi Arabia have revealed a tremendous increase in its prevalence among children over the last few decades. A systematic review examined the national prevalence of caries among Saudi schoolchildren from 1988 to 2010. The review revealed that dental caries is highly prevalent across Saudi Arabia, particularly in Riyadh City. The caries prevalence in primary teeth was approximately 80% with a mean dmft of 5.0, while in permanent teeth, the prevalence was estimated to be 70% with a mean DMF value of 3.5. A recent systematic review evaluated caries prevalence from 1999 to 2019. The results showed that the proportion level for caries among schoolchildren is high, ranging from 0.21 to 1.00 for primary teeth and from 0.05 to 0.99 for permanent teeth. This emphasises that dental caries remains a significant oral health issue in Saudi Arabia.

In Riyadh city, several studies have consistently indicated a high prevalence of dental caries and DMFT values in children. A national study explored caries prevalence and severity among schoolchildren across Saudi Arabia. This study included a nationwide sample of 19,870 school students. The study found that 65.6% of examined children had caries, with a mean dmft of 3.93 ± 3.60 and a mean DMFT of 2.42 ± 2.52. It was observed that Riyadh City exhibited the highest rate of missing teeth at 10.2%. Despite the lower prevalence of caries reported in this study compared to previous studies, it remained higher than that reported in other countries, such as the United Kingdom, with a caries prevalence of 29.3% among 5-year-old children. This illustrates that caries continues to be a significant concern and the primary oral health issue among Saudi children.

Implementation of oral health programmes in school settings is considered one of the most effective approaches for improving children's oral health, as they can reach many schoolchildren. The report titled "Oral Health Promotion: An Essential Element of a Health-Promoting School" recognised schools as an ideal environment for promoting oral health due to their significant impact on children's oral health status, knowledge, and behaviours. The report shed light on global evidence supporting the efficacy of oral health programmes in schools. It was noticed that countries adopting public health programmes, including school-based oral health programmes, have witnessed a reduction in caries prevalence.

On the other hand, the caries prevalence in Saudi Arabia remains high. Over the years, the Saudi Ministry of Health has been active in promoting oral health and has implemented a range of oral health programmes to enhance oral health, control and prevent oral diseases, including dental caries. However, no consistent national oral health school-based programmes are implemented in Saudi Arabia.

There is strong and sufficient evidence regarding the effectiveness of supervised toothbrushing with fluoride toothpaste on the oral health status of preschool and school children. A study evaluated evidence-based oral health promotion programmes. The findings indicated that supervised toothbrushing interventions have resulted in caries reductions of 40%. The author also reported that supervised toothbrushing interventions are cost-effective and more efficient when specifically targeted towards high-risk populations. The programmes that had the strongest evidence for preventing caries were implemented in Scotland, England, and Jordan. The study in Jordan, a country with a similar cultural background and social norms to Saudi Arabia. The programme lasted four years and involved daily supervised toothbrushing at school. The results showed that children in the supervised toothbrushing group exhibited better caries status and were up to 6 times less likely to have caries than the control group.

A systematic review concluded that the effectiveness and benefits of using fluoridated toothpaste to prevent dental caries among children are well established. Research indicates that dental caries in primary dentition can progress rapidly over one year. Another systematic review revealed that 3.8% to 12.2% of children develop cavities in their primary teeth annually. The rapid progression of caries in primary teeth within a year, especially when using the WHO criteria that records only cavitated lesions, emphasises the importance of early detection and preventive measures to manage caries in primary dentition effectively. It is also worth noting that this quick progression of caries in the primary teeth will allow detection of changes in caries within one year. Supervised toothbrushing with fluoridated toothpaste can be effective in reducing this risk, as it helps in the early management of incipient caries, preventing their progression to cavitated lesions.

A systematic review to evaluate the effectiveness of oral health promotion interventions among children found that interventions that include supervised toothbrushing with fluoridated toothpaste were more effective in preventing caries in primary teeth. Another review explored a range of school-based supervised toothbrushing programmes, concluding that children participating in toothbrushing interventions are most likely to have better oral hygiene practices, oral cleanliness, and gingival health.

To date, no supervised toothbrushing programmes have been implemented in school settings in Saudi Arabia. Given the robust evidence of supervised toothbrushing and the high risk of dental caries among Saudi children, implementing this programme is expected to be an effective strategy for reducing caries.

The evidence for the effectiveness of school-based oral health education programmes indicates that they yield positive outcomes for children's knowledge acquisition. There is some evidence on the effectiveness of integrating preschool and school-based supervised toothbrushing programmes with oral health education. A systematic review comprised four randomised controlled trials. Interventions included oral health education and supervised toothbrushing sessions. The authors reported limited evidence of these interventions on caries prevention; however, it was noted that they have a positive impact on plaque levels and children's knowledge. Three studies found a statistically significant reduction in plaque in the intervention groups compared to the control groups.

According to a recent systematic review, oral health education sessions incorporated lectures, audiovisual aids, and activities effectively reduced plaque and bleeding scores, and enhanced the knowledge and behaviour of schoolchildren aged 6 to 12. Another recent systematic review showed that the oral health education interventions, such as oral health education "lectures, albums, slides, leaflets, counselling, games, drawings, theatre, dieting guidance, toothbrushing instructions, toothbrushing demonstration with models, and supervised toothbrushing, were significantly effective on schoolchildren's oral health status.

A randomised controlled trial was conducted in 2022 to evaluate the effectiveness of oral health promotion programmes among 702 primary students in Sakaka, Saudi Arabia. The study demonstrated a significant reduction in dental caries, indicating that oral health education involving teachers with reinforcement sessions is an effective approach for improving the oral health of Saudi children. In addition, another study found that oral health education programmes in primary schools in Riyadh, Saudi Arabia, positively impacted students' oral health knowledge and behaviours. Based on the previous evidence, oral health education sessions involving teachers may be applicable and effective for the Saudi population.

Limited research has been conducted into the practical implementation of supervised toothbrushing programmes. A pilot study evaluated the feasibility of implementing preventive programmes, including fluoride varnish and toothbrushing programmes, among 3 to 7-year-old students in primary schools in London, UK. The findings showed that the toothbrushing programme was feasible to execute in schools and was accepted by all stakeholders, including parents, school staff and dental teams. The study discovered that appointing school staff in each school to lead the programme and facilitate communication contributes to its successful implementation. A recent pilot study examined the feasibility of conducting supervised toothbrushing and fluoride varnish programmes and their effects on dental caries in Derby City, England. The results indicated a decrease in dental caries and improvement in oral hygiene and dental attendance. Frequently reported Facilitators to supervised toothbrushing implementation include programme flexibility, school staff positive attitudes, community volunteer involvement, and the development of toothbrushing habits. In the context of Saudi Arabia, the majority of participating teachers expressed interest in oral health education programmes and supported their inclusion in the curriculum.

Rationale for the study The high prevalence of caries in Saudi Arabia and its impact on general health make it increasingly important to establish effective preventive oral health measures. The WHO recommended conducting oral health programmes to improve children's oral health in school settings. Unfortunately, most Saudi children are at high risk for dental caries. Even with the nationwide oral health programmes aimed at caries prevention among schoolchildren and free oral healthcare, the caries prevalence remains high. No consistent national oral health school-based promotion programmes have been implemented in Saudi Arabia. From 1993 to 2018, the Ministry of Health has been implementing various school-based oral health programmes. However, no research determines the extent of the changes that have occurred, nor has it evaluated the feasibility, facilitators, barriers, impact, or outcomes of these programmes. Furthermore, none of the programmes included a supervised toothbrushing intervention. Therefore, this study aims to address this research gap by assessing the feasibility of implementing supervised toothbrushing and oral health education programmes, as well as identifying the facilitators and barriers to implementation. While supervised toothbrushing has proven effective in other countries, it remains unclear whether such a programme is transferable and acceptable within the Saudi context. The study specifically seeks to determine the acceptability of the programme among teachers and students, assess willingness to participate among children and their parents, and explore the capacity of schoolteachers to supervise daily toothbrushing sessions. To enhance the oral health of Saudi children, it is important to assess which of the oral health programmes are needed and applicable to the Saudi community, as well as determine the best approach for implementation. Promoting oral health through evidence-based programmes in primary schools may be highly correlated with improving oral health outcomes for this population and acquiring behaviours that are crucial to maintaining optimal oral health throughout life.

Aim and Objectives

The objectives are:

1. To assess the feasibility of implementing supervised toothbrushing and oral health education programmes in primary schools in Riyadh, Saudi Arabia
2. To identify facilitators and barriers to the implementation, focusing on the programme acceptance, school staff participation, and adherence to the supervision guide
3. To determine the impact of programmes on students' self-reported oral health status, risk behaviour, and quality of life
4. To examine the impact of the programmes on plaque and gingival health status
5. To evaluate the impact of the programmes on dental caries incidence

ELIGIBILITY:
Inclusion Criteria:

* Students aged 5 to 8 years are in the first grade of primary school.
* Students must be medically fit.
* Students who provide consent to participate in the study.
* Students for whom a parent/ legal guardian has signed the consent form.

Exclusion Criteria:

* Students with systemic disease or any medically compromised condition that hinders their participation in the programme.
* Students who refuse to provide consent to participate in the study.
* Students for whom a parent/ legal guardian has refused to sign the consent form.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Estimated)
Dates: Start 2024-08-18 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of implementing supervised toothbrushing and oral health education programmes based on qualitative interviews | At the end of the academic year (approximately 9 to 12 months after programme initiation)
  Feasibility will be assessed through semi-structured interviews conducted with school staff and dental professionals. The interviews will explore programme acceptability, staff engagement, adherence to toothbrushing supervision protocols, and perceived barriers and facilitators to implementation. Data will be thematically analysed to identify factors influencing the programme implemation.

SECONDARY OUTCOMES:
Change in dental caries prevalence using dmft score | Baseline and one-year follow-up
  Dental examinations will be conducted at baseline and follow-up after one academic year. Dental caries will be assessed using the decayed, missing, and filled teeth (dmft) index for primary teeth and DMFT index for permanent teeth. The dmft/DMFT score represents the total number of teeth that are decayed (d/D), missing due to caries (m/M), or filled (f/F). A higher score indicates greater caries experienceChange over time will be analysed using appropriate statistical methods (e.g., odds ratios with 95% confidence intervals)
Change in plaque and gingival health using Modified Plaque and Bleeding Scores | Baseline, 9 months, and 12 months after programme initiation
  Oral hygiene and gingival health will be assessed on six Ramfjord teeth using the Modified Plaque Score (MPS) and Modified Bleeding Score (MBS). The MPS evaluates plaque accumulation on tooth surfaces, scored from 0 (no plaque visible, even after probing) to 2 (visible plaque without probing), with results expressed as a percentage plaque score. The MBS assesses gingival bleeding on probing, scored as 0 (no bleeding) or 1 (presence of marginal bleeding within 30 seconds), also expressed as a percentage bleeding score. These scores will be used to monitor changes in plaque levels and gingival inflammation over time. Assessments will be conducted at baseline, 9 months, and 12 months after programme initiation.
Children's oral health status, behaviours, risk factors, quality of life, and socio-demographic factors using the WHO Oral Health Questionnaire for Children | Baseline and one-year follow-up
  The World Health Organisation's Oral Health Questionnaire for Children (WHO, 2013) will be used to assess multiple domains, including oral health status, oral health-related behaviours, risk factors, quality of life related to oral health, and relevant socio-demographic information.

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical considerations related to the confidentiality of minor participants. Only aggregated and anonymised results will be published.

REFERENCES:
- [Background] Alshammari FR, Alamri H, Aljohani M, Sabbah W, O'Malley L, Glenny AM. Dental caries in Saudi Arabia: A systematic review. J Taibah Univ Med Sci. 2021 Jul 22;16(5):643-656. doi: 10.1016/j.jtumed.2021.06.008. eCollection 2021 Oct. PMID 34690643
- [Background] Aljanakh M, Siddiqui AA, Mirza AJ. Teachers' knowledge about oral health and their interest in oral health education in Hail, Saudi Arabia. Int J Health Sci (Qassim). 2016 Jan;10(1):87-93. PMID 27004061
- [Background] Cooper AM, O'Malley LA, Elison SN, Armstrong R, Burnside G, Adair P, Dugdill L, Pine C. Primary school-based behavioural interventions for preventing caries. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD009378. doi: 10.1002/14651858.CD009378.pub2. PMID 23728691
- [Background] Wang MC, Marshman Z, Chen WH, Shih WY. A qualitative study of barriers and facilitators to the implementation of a pilot school-based, toothbrushing programme. BMC Oral Health. 2022 Oct 24;22(1):451. doi: 10.1186/s12903-022-02494-7. PMID 36280822
- [Background] Tickotsky N, Petel R, Araki R, Moskovitz M. Caries Progression Rate in Primary Teeth: A Retrospective Study. J Clin Pediatr Dent. 2017;41(5):358-361. doi: 10.17796/1053-4628-41.5.358. PMID 28872992
- [Background] Stein C, Santos NML, Hilgert JB, Hugo FN. Effectiveness of oral health education on oral hygiene and dental caries in schoolchildren: Systematic review and meta-analysis. Community Dent Oral Epidemiol. 2018 Feb;46(1):30-37. doi: 10.1111/cdoe.12325. Epub 2017 Aug 16. PMID 28815661
- [Background] Orfali SM, Alrumikhan AS, Assal NA, Alrusayes AM, Natto ZS. Prevalence and severity of dental caries in school children in Saudi Arabia: A nationwide cross-sectional study. Saudi Dent J. 2023 Dec;35(8):969-974. doi: 10.1016/j.sdentj.2023.09.008. Epub 2023 Sep 22. PMID 38107051
- [Background] Marinho VC, Higgins JP, Sheiham A, Logan S. Fluoride toothpastes for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2003;2003(1):CD002278. doi: 10.1002/14651858.CD002278. PMID 12535435
- [Background] Hummel R, Akveld NAE, Bruers JJM, van der Sanden WJM, Su N, van der Heijden GJMG. Caries Progression Rates Revisited: A Systematic Review. J Dent Res. 2019 Jul;98(7):746-754. doi: 10.1177/0022034519847953. Epub 2019 May 9. PMID 31070943
- [Background] Halawany HS, Al Badr A, Al Sadhan S, Al Balkhi M, Al-Maflehi N, Abraham NB, Jacob V, Al Sherif G. Effectiveness of oral health education intervention among female primary school children in Riyadh, Saudi Arabia. Saudi Dent J. 2018 Jul;30(3):190-196. doi: 10.1016/j.sdentj.2018.04.001. Epub 2018 May 4. PMID 29942102
- [Background] Gray-Burrows KA, Day PF, El-Yousfi S, Lloyd E, Hudson K, Marshman Z. A national survey of supervised toothbrushing programmes in England. Br Dent J. 2023 Aug 21. doi: 10.1038/s41415-023-6182-1. Online ahead of print. PMID 37604921
- [Background] Geetha Priya PR, Asokan S, Janani RG, Kandaswamy D. Effectiveness of school dental health education on the oral health status and knowledge of children: A systematic review. Indian J Dent Res. 2019 May-Jun;30(3):437-449. doi: 10.4103/ijdr.IJDR_805_18. PMID 31397422
- [Background] Dickson-Swift V, Kenny A, Gussy M, de Silva AM, Farmer J, Bracksley-O'Grady S. Supervised toothbrushing programs in primary schools and early childhood settings: A scoping review. Community Dent Health. 2017 Dec 1;34(4):208-225. doi: 10.1922/CDH_4057Dickson-Swift18. PMID 29119741
- [Background] de Silva AM, Hegde S, Akudo Nwagbara B, Calache H, Gussy MG, Nasser M, Morrice HR, Riggs E, Leong PM, Meyenn LK, Yousefi-Nooraie R. Community-based population-level interventions for promoting child oral health. Cochrane Database Syst Rev. 2016 Sep 15;9(9):CD009837. doi: 10.1002/14651858.CD009837.pub2. PMID 27629283
- [Background] Chandio N, Micheal S, Tadakmadla SK, Sohn W, Cartwright S, White R, Sanagavarapu P, Parmar JS, Arora A. Barriers and enablers in the implementation and sustainability of toothbrushing programs in early childhood settings and primary schools: a systematic review. BMC Oral Health. 2022 Jun 18;22(1):242. doi: 10.1186/s12903-022-02270-7. PMID 35717199
- [Background] Burgess-Allen J, Braithwaite M, Whiston S. Challenges associated with implementation of a school-based tooth-brushing and fluoride varnish programme in a diverse and transient urban population. Community Dent Health. 2018 May 30;35(2):71-74. doi: 10.1922/CDH_4101Burgess-Allen04. PMID 29558062
- [Background] Alkarimi HA, Watt RG, Pikhart H, Sheiham A, Tsakos G. Dental caries and growth in school-age children. Pediatrics. 2014 Mar;133(3):e616-23. doi: 10.1542/peds.2013-0846. Epub 2014 Feb 17. PMID 24534405
- [Background] Alhabdan YA, Albeshr AG, Yenugadhati N, Jradi H. Prevalence of dental caries and associated factors among primary school children: a population-based cross-sectional study in Riyadh, Saudi Arabia. Environ Health Prev Med. 2018 Nov 30;23(1):60. doi: 10.1186/s12199-018-0750-z. PMID 30497366
- [Background] Alwayli HM, Alshiha SA, Alfraih YK, Hattan MA, Alamri AA, Aldossary MS. A survey of fissure sealants and dental caries prevalence in the first permanent molars among primary school girls in Riyadh, Saudi Arabia. Eur J Dent. 2017 Oct-Dec;11(4):455-460. doi: 10.4103/ejd.ejd_189_17. PMID 29279670
- [Background] Al-Malik MI, Rehbini YA. Prevalence of dental caries, severity, and pattern in age 6 to 7-year-old children in a selected community in Saudi Arabia. J Contemp Dent Pract. 2006 May 1;7(2):46-54. PMID 16685294
- [Background] Al-Jundi SH, Hammad M, Alwaeli H. The efficacy of a school-based caries preventive program: a 4-year study. Int J Dent Hyg. 2006 Feb;4(1):30-4. doi: 10.1111/j.1601-5037.2006.00156.x. PMID 16451437
- [Background] Al Agili DE. A systematic review of population-based dental caries studies among children in Saudi Arabia. Saudi Dent J. 2013 Jan;25(1):3-11. doi: 10.1016/j.sdentj.2012.10.002. Epub 2012 Nov 10. PMID 23960549
- See also: Related Info — https://www.researchgate.net/publication/273441571_Are_the_Approximal_Caries_Lesions_in_Primary_Teeth_a_Challenge_to_Deal_With_-_A_Critical_Appraisal_of_Recent_Evidences_in_This_Field
- See also: Related Info — https://www.moh.gov.sa/en/Ministry/Projects/tooth-decay/Pages/default.aspx
- See also: Related Info — https://www.gov.uk/government/statistics/oral-health-survey-of-5-year-old-children-2022/national-dental-epidemiology-programme-ndep-for-england-oral-health-survey-of-5-year-old-children-2022
- See also: Related Info — https://assets.publishing.service.gov.uk/media/5a7d6f6bed915d269ba8aa6a/CBOHMaindocumentJUNE2014.pdf
- See also: Related Info — https://content.health.vic.gov.au/sites/default/files/migrated/files/collections/policies-and-guidelines/f/final-oral-health-resource-may-2011-web-version---pdf.pdf
- See also: Related Info — https://iris.who.int/bitstream/handle/10665/70207/WHO_NMH_NPH_ORH_School_03.3_eng.pdf?sequence=1&isAllowed=y
- See also: Related Info — https://www.who.int/publications/i/item/9789240061484